CLINICAL TRIAL: NCT02830854
Title: Molecular Hydrogen for Cognitive Function and Performance in Elderly
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Novi Sad, Faculty of Sport and Physical Education (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: DK-DR16-02
Record Dates: First submitted 2016-07-07; First posted 2016-07-13 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Cognitive Impairments; Aging
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Hydrogen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Molecular Hydrogen (Experimental): Molecular hydrogen: 20 min per day of 3% H2 during 4 weeks
  Interventions: Other: Molecular Hydrogen

INTERVENTIONS:
Other: Molecular Hydrogen

SUMMARY:
A variety of non-pharmacological interventions have been used in the management of Alzheimer's disease (AD) and similar cognitive disorders in elderly, yet no therapeutic modality has demonstrated conclusive positive results in terms of effectiveness. Although it is still unknown what triggers AD, recent studies have shown that AD is associated with brain energy depletion, oxidative stress, and mitochondrial dysfunction. Since supplemental molecular hydrogen (H2) supports cell energy production and acts as a highly bioavailable mitochondria-related antioxidant, it may provide an ideal agent to facilitate treatment and perhaps prevention of AD and similar cognitive disorders in elderly. The overall hypothesis to be evaluated in this project is that administration of H2 will positively affect patient-reported outcomes and clinical biomarkers in men and women suffering from AD.

ELIGIBILITY:
Inclusion Criteria:

* Age over 65
* No psychiatric comorbidities

Exclusion Criteria:

* Use of dietary supplements 4 weeks before study commence

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 13 (Actual)
Dates: Start 2016-07; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
ADAS-Cog score for cognitive function | Change from Baseline ADAS-Cog Score at 4 weeks
  ADAS-Cog total score and scores for 4 separate cognitive domains (memory, orientation, praxis, and language) will be evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Applied Bioenergetics Lab at Faculty of Sport and PE, Novi Sad, Vojvodina, Serbia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ostojic SM. Molecular hydrogen: An inert gas turns clinically effective. Ann Med. 2015 Jun;47(4):301-4. doi: 10.3109/07853890.2015.1034765. Epub 2015 May 4. PMID 25936365
- [Background] Ostojic SM. Targeting molecular hydrogen to mitochondria: barriers and gateways. Pharmacol Res. 2015 Apr;94:51-3. doi: 10.1016/j.phrs.2015.02.004. Epub 2015 Feb 24. PMID 25720951
- [Background] Ohno K, Ito M, Ichihara M, Ito M. Molecular hydrogen as an emerging therapeutic medical gas for neurodegenerative and other diseases. Oxid Med Cell Longev. 2012;2012:353152. doi: 10.1155/2012/353152. Epub 2012 Jun 8. PMID 22720117